

## UNDERTAKING FORM FOR RESEARCHERS CONDUCTING OR PARTICIPATING IN RESEARCH AT UÜ-SK

| Dok.Kodu | : FR-HYH-23 | İlk Yay.Tarihi | : 04 Ocak 2011 | Sayfa<br>1 / 1 |
|----------|-------------|----------------|------------------|----------------|
| Rev. No | : 01 | Rev.Tarihi | : 19 Aralık 2011 | |

As the principal investigators and co-investigators who participated in the study titled "The Role and Limitations of Ultrasound Use for Decannulation; A Prospective Observational Study," the undersigned; 1. I declare that the information provided in the application is accurate and that I will comply with national and international regulations and fulfill their requirements throughout the research.

- 2. I will inform the research team about the research.
- 3. I will also verbally inform the volunteers when obtaining "Informed Consent" (Informed Voluntary Consent) from patients and/or healthy volunteers.
- 4. I will not perform any procedures on the volunteers other than those specified in the "Informed Consent" (Informed Voluntary Consent) form.
- 5. I will not use the information and materials obtained from the volunteers for purposes other than those specified in the research protocol.
- 6. I will provide a copy of the "Informed Consent" (Informed Voluntary Consent) forms to the volunteers.
- 7. I will keep a copy of the "Informed Consent" (Informed Voluntary Consent) forms obtained from inpatient volunteers in the "consents" separator in the patient file. I will place it under the "Informed Consent" form obtained from outpatient clinic patients and healthy volunteers using electronic patient files.

I/we declare and undertake that I will keep a copy of the "Informed Consent" form in the study file.

- 9. I will notify the Uludağ University Faculty of Medicine Clinical Research Ethics Committee in a timely manner, in accordance with the principle of confidentiality, of the exact start date of the study after ethical approval is obtained, any changes made to the study, and the names and protocol numbers of the volunteers included in the study.
- 10. I will submit a copy of the final report to the Uludağ University Faculty of Medicine Clinical Research Ethics Committee within one (1) year after the study is concluded.

Date: 26/06/2024